CLINICAL TRIAL: NCT04915131
Title: A Cross-sectional, Interventional, Single-arm Clinical Study for Validating the Equivalence of Bloomlife MFM-Pro to Clinical Standard-of-care for Fetal Heart Rate and Maternal Heart Rate When Performing Antepartum Fetal Monitoring
Brief Title: A Clinical Study for Validating the Equivalence of Bloomlife MFM-Pro to Clinical Standard-of-care for Performing Antepartum Fetal Monitoring
Acronym: NST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bloom Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NST-01-2021-US
Record Dates: First submitted 2021-04-10; First posted 2021-06-07 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Fetal Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Bloomlife MFM-Pro (Other)
  Interventions: Device: Bloomlife MFM-Pro

INTERVENTIONS:
Device: Bloomlife MFM-Pro — Bloomlife MFM-Pro is a non-invasive, wireless, external monitoring system used to measure fetal heart rate and maternal heart rate on pregnant women with a singleton pregnancy.
  The system acquires biopotential signals from abdominal surface electrodes.

SUMMARY:
Bloomlife MFM-Pro is a non-invasive, wireless, external monitoring system used to measure fetal heart rate and maternal heart rate on pregnant women with a singleton pregnancy, starting from 32 weeks of gestation.

The purpose of this study is to validate that the Bloomlife MFM-Pro is equivalent to clinical standard-of-care for fetal heart rate and maternal heart rate when performing antepartum fetal monitoring.

DETAILED DESCRIPTION:
The study consisted of 2 phases: a pilot phase and a pivotal phase. The pilot phase of the study was aimed at testing the Bloomlife MFM-Pro device prior to validation in the pivotal phase of the study. The pivotal phase of the study was aimed at validating that the Bloomlife MFM-Pro is equivalent to clinical standard-of-care for fetal heart rate and maternal heart rate when performing antepartum fetal monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman ≥ 18 years old
* Gestational age ≥ 32 weeks and 0 days
* Singleton pregnancy
* Ability to read and understand English or Spanish
* Willingness to participate in the study

Exclusion Criteria:

* Implanted pacemaker or any other implanted electrical device
* Plurality higher than 1
* History of allergies to skin adhesives
* Irritated or lesioned skin at the Bloomlife MFM-Pro electrodes locations
* Contraindication to the use of CTG

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avinash Patil, Principal Investigator — Valley Perinatal Services
Locations (2):
- United States (2):
  - Valley Perinatal Services, Phoenix, Arizona
  - Ochsner, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Bloomlife MFM-Pro, Pilot Phase: The pilot phase of the study was aimed at testing the Bloomlife MFM-Pro device prior to validation in the pivotal phase of the study.
- Bloomlife MFM-Pro, Pivotal Phase: The pivotal phase of the study was aimed at validating that the Bloomlife MFM-Pro is equivalent to clinical standard-of-care for fetal heart rate and maternal heart rate when performing antepartum fetal monitoring.
Period: Overall Study
Arm/Group | Bloomlife MFM-Pro, Pilot Phase | Bloomlife MFM-Pro, Pivotal Phase
Started | 60 (Participants enrolled in the pilot phase of the study) | 61 (Participants enrolled in the pivotal phase of the study)
Analysis Population | 54 (The Analysis Population includes all enrolled participants without major protocol deviation or technical failure. 4 participants were excluded from the analysis due to protocol deviation. 2 participants were excluded from the analysis due to technical failures of the clinical tools.) | 56 (The Analysis Population includes all enrolled participants without major protocol deviation or technical failure. 5 participants were excluded from the analysis due to protocol deviation.)
Completed | 60 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bloomlife MFM-Pro, Pilot Phase | Bloomlife MFM-Pro, Pivotal Phase | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (6.31) | 30.4 (5.69) | 30.1 (6.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 61 | 121
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 19 | 43
  Not Hispanic or Latino | 36 | 40 | 76
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 13 | 13 | 26
  White | 31 | 30 | 61
  More than one race | 8 | 10 | 18
  Unknown or Not Reported | 1 | 2 | 3
Pre-pregnancy Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.7 (7.81) | 33.19 (7.776) | 31.96 (7.89)
Gestational Age [Mean (Standard Deviation); unit: weeks] | 35.8 (1.96) | 35.51 (2.102) | 35.65 (2.04)

OUTCOME MEASURES:

1. Primary Outcome: Extent of Agreement Between Bloomlife MFM-Pro and CTG in Fetal Heart Rate
Time Frame: 5 minutes
Population: The Analysis Population includes all enrolled patients without major protocol deviations or technical failure
Measure: Mean (95% Confidence Interval); unit: BPM
Groups:
- Bloomlife MFM-Pro, Pivotal Phase: The pivotal phase of the study was aimed at validating that the Bloomlife MFM-Pro is equivalent to clinical standard-of-care for fetal heart rate and maternal heart rate when performing antepartum fetal monitoring."
Arm/Group | Bloomlife MFM-Pro, Pilot Phase | Bloomlife MFM-Pro, Pivotal Phase
Number analyzed (Participants) | 54 | 56
BPM
  Lower Limit of Agreement | -5.46 [-5.57 to -5.36] | -5.57 [-6.92 to -4.16]
  Upper Limit of Agreement | 6.04 [5.93 to 6.14] | 6.04 [4.75 to 7.27]

2. Primary Outcome: Extent of Agreement Between Bloomlife MFM-Pro and CTG in Maternal Heart Rate
Time Frame: 5 minutes
Population: Analysis Population includes all enrolled patients without major protocol deviation or technical failure.
Measure: Mean (95% Confidence Interval); unit: BPM
Arm/Group | Bloomlife MFM-Pro, Pilot Phase | Bloomlife MFM-Pro, Pivotal Phase
Number analyzed (Participants) | 54 | 56
BPM
  Lower Limit of Agreement | -2.27 [-2.51 to -2.03] | -1.84 [-2.05 to -1.66]
  Upper Limit of Agreement | 3.56 [3.32 to 3.80] | 2.67 [2.38 to 2.98]

ADVERSE EVENTS:
Time Frame: Measurement time + 7-day follow-up period
Description: Bloomlife MFM-Pro is a safe, non-invasive device that measures standard physiological parameters. Risk assessment and management was performed in compliance with ISO 14791 standard. The anticipated adverse device effects involved with the use of the device include skin irritations and sensitization, which is considered a minor physical risks directly related to the use of Bloomlife MFM-Pro. The risk of mortality and serious adverse events is considered negligible.
Arm/Group | Bloomlife MFM-Pro, Pilot Phase | Bloomlife MFM-Pro, Pivotal Phase
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 1/60 | 1/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bloomlife MFM-Pro, Pilot Phase (N=60) | Bloomlife MFM-Pro, Pivotal Phase (N=61)
Discomfort at electrode location (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Irritation between two measurement electrodes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT04915131/Prot_SAP_000.pdf